CLINICAL TRIAL: NCT00425789
Title: Hyperbaric Therapy and Healing From Deep Chemical Peel
Brief Title: Hyperbaric Therapy and Deep Chemical Peeling
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 115/05
Record Dates: First submitted 2007-01-22; First posted 2007-01-23 (Estimated); Last update posted 2011-04-05 (Estimated); Status verified 2005-12

CONDITIONS: Chemical Peeling
Keywords: Deep Chemical Peeling; Hyperbaric Therapy; post-deep peel
MeSH Terms: interventions — Therapeutics

INTERVENTIONS:
Procedure: Treatment with Hyperbaric oxygen

SUMMARY:
To evaluate whether treatment with Hyperbaric oxygen can accelerate skin recovery after deep peeling, and decrease frequency and severity of local side effects and complications.

20 post peel patients will recieve 5 daily hyperbaric treatments, starting from day 7 to peel.Patient's followup will include self- filling questionnaire and photographs

DETAILED DESCRIPTION:
The study will include 40 post-deep peel women (exoderm), older than 18 years old, treated by the same dermatologist.

The treatment group will recieve 5 consecutive daily hyperbaric treatments, 1 hours long each, at 2 ATF, starting from day 7 to peel. Prior to treatment, each patient will be signed on informed consent and will have complete physical examination.

The control group will be matched by the following parameters: age, skin color and type, and indication for peeling, and will be picked up by the dermatologist.

Patients will be excluded if they have known middle ear disease, chronic lung disease or claustrophobia.

Follow -up:

The same dermatologist will follow-up, on regular dates: the follow-up examination will start at day 1 to mask\occlusive dressing removal (equivalent to day 7 post-peel), and at days 7, 28, and after 3 months. All follow-up examinations will take place at noon (04-08 pm) regularly.

Efficacy parameters:

All patients will be asked to fill up a daily questionnaire on the first week after peel, and score the severity of pain, pruritus and tightness of facial skin (1 to 5). They will also mention the daily analgesic usage.

Parameters that will be evaluated by the dermatologist during the study will be: tightness of the skin, pain/burning, pruritus/stinging, swelling/edema, erythema, crusting, and scaling, assessed on a 4-point severity scale (0- best, 3- worst).

Photographs:

Photographs of the patients in 5 angles views will be taken on the day of peel, day of mask removal (7), day 28 and after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* The study will include 40 post-deep peel women (exoderm), older than 18 years old, treated by the same dermatologist (dr. Landau).
* The treatment group will receive 5 consecutive daily hyperbaric treatments, 1 hours long each, at 2 ATF, starting from day 7 to peel. Prior to treatment, each patient will be signed on informed consent and will have complete physical examination.
* The control group will be matched by the following parameters: age, skin color and type, and indication for peeling, and will be picked up by the dermatologist.

Exclusion Criteria:

* Patients will be excluded if they have known middle ear disease, chronic lung disease or claustrophobia

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-01; Study Completion 2007-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tal Friedman, MD, Principal Investigator — Assaf-Harofeh Medical Center; Shai Efrati, MD, Study Director — Assaf-Harofeh Medical Center
Locations (1):
- Research & Development Unit, Assaf-Harofeh Medical Center, Ẕerifin, Israel